CLINICAL TRIAL: NCT03812302
Title: Evaluating the Use of Gallium-68 HA-DOTATATE Positron Emission Tomography/Computerized Tomography (PET/CT) in Patients With Giant Cell Arteritis (GCA.)
Brief Title: Use of Gallium-68 HA-DOTATATE PET/CT in Giant Cell Arteritis (GCA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00085448
Record Dates: First submitted 2019-01-18; First posted 2019-01-23 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Giant Cell Arteritis
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Intervention Model Description: 68-Ga HA-DOTATATE PET/CT will be performed in all participants as part of study protocol. Participants will receive an intravenous infusion of 3MBq/kg of 68Ga HA-DOTATATE (to max 200 MBq), followed by CT and PET imaging 60 minutes later. Tracer uptake in each vascular territory will be interpreted qualitatively and quantitatively.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DOTATATE (Experimental): All 15 GCA patients will undergo 68-Ga HA-DOTATATE PET/CT imaging at baseline, in addition to FDG PET/CTA (as part of standard of care). DOTATATE PET/CT imaging will be repeated at 6 months follow-up.
  Interventions: Diagnostic Test: 68-Ga HA-DOTATATE PET/CT

INTERVENTIONS:
Diagnostic Test: 68-Ga HA-DOTATATE PET/CT — See arm description.

SUMMARY:
The aim of this study is to compare the use of FDG PET/CT to Ga-68 HA-DOTATATE (abbreviated DOTATATE) PET/CT in patients with active giant cell arteritis (GCA) started on prednisone to understand if DOTATATE can identify more areas of active blood vessel inflammation than FDG.

DETAILED DESCRIPTION:
The aim of this study is to prospectively evaluate the potential use of 68-Ga HA-DOTATATE PET/CT for detecting medium-large vessel inflammation in a small number of GCA patients with active disease, as compared to FDG PET/CT, and to understand if DOTATATE uptake correlates with disease activity. Fifteen patients with active GCA (either newly-diagnosed or recently relapsed disease) who are receiving glucocorticoids will be enrolled. Participants will undergo baseline FDG PET/CT and baseline DOTATATE PET/CT scan. Tracer uptake will be described in 8 major vascular territories. DOTATATE PET/CT will be repeated again in 6 months, and tracer uptake will be correlated to clinical disease activity, and medication use.

ELIGIBILITY:
Inclusion Criteria:

Participants must:

1. Meet the revised GCA diagnosis criteria (modified from ref 1)
2. Have either newly-diagnosed or relapsing disease
3. Have active disease (modified from ref 1, to remove ESR/CRP requirements)
4. Have been empirically started on glucocorticoid treatment (or had baseline glucocorticoid dose increased, in the case of relapsers) ≤ 2 weeks of enrolment
5. Participant must be have had (or will be willing to undergo) an urgent FDG-PET/CT as part of routine clinical care.

GCA diagnosis criteria (modified from ref 1, to remove ESR requirement).

1. Age ≥ 50 years
2. And at least 1 of a. or b. :

   1. Unequivocal cranial symptoms of GCA (new headache, scalp or temporal artery tenderness, ischemia-related vision loss, jaw/mouth claudication
   2. Unequivocal symptoms of polymyalgia rheumatica (PMR), defined as shoulder and/or hip girdle pain associated with inflammatory stiffness
3. And at least 1 of a. or b.:

   1. Temporal artery biopsy revealing features of GCA
   2. Evidence of large-vessel vasculitis by angiography or cross-sectional imaging study such as magnetic resonance angiography (MRA), computed tomography angiography (CTA), or positron emission tomography-computed tomography (PET-CT)

Exclusion Criteria:

* Patients not meeting the above criteria or who are unable to provide informed consent will be excluded.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison of FDG vs DOTATATE vascular uptake in individual vascular territories using target-blood pool ratios (TBR) | time 0 (baseline)

SECONDARY OUTCOMES:
Qualitative comparison of FDG vs DOTATATE vascular uptake in individual vascular (scores 0-3) territories using visual uptake scores | time 0 (baseline)
Changes in vascular DOTATATE uptake scores over time (quantitatively and qualitatively) | 6 months
Correlation between vascular DOTATATE uptake scores and clinical status | 0 and 6 months
Correlation between vascular DOTATATE uptake scores and cumulative glucocorticoid exposure | 0 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Alison Clifford, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Unizony SH, Dasgupta B, Fisheleva E, Rowell L, Schett G, Spiera R, Zwerina J, Harari O, Stone JH. Design of the tocilizumab in giant cell arteritis trial. Int J Rheumatol. 2013;2013:912562. doi: 10.1155/2013/912562. Epub 2013 Apr 7. PMID 23653652
- [Derived] Clifford AH, Abele J, Hung R, Wuest F, Andersson J, Pike S, Yacyshyn E, Lenza E, Jickling G, Raggi P, Cohen Tervaert JW. Comparison of [18F]fluorodeoxyglucose and [68Ga]Gallium DOTA-TATE in patients with active giant cell arteritis. EJNMMI Rep. 2025 Mar 1;9(1):7. doi: 10.1186/s41824-025-00242-y. PMID 40021570